CLINICAL TRIAL: NCT06145386
Title: "The Effect of Aerobic Exercise and Strength Training on Physical Activity Level, Quality of Life and Anxiety-Stress Disorder in Young Adults With and Without Covid-19"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ozge Mine Yilmaz, PhD Student, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pamukkale Universityy
Record Dates: First submitted 2023-11-22; First posted 2023-11-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: aerobic exercise, strength training, pulmonary capacity
MeSH Terms: conditions — COVID-19 | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 positive (Experimental)
  Interventions: Behavioral: Aerobic Exercise and Strength Training
- COVID-19 negative (Experimental)
  Interventions: Behavioral: Aerobic Exercise and Strength Training

INTERVENTIONS:
Behavioral: Aerobic Exercise and Strength Training — Aerobic Exercise and Strength Training on Physical Activity Level, Quality of Life and Anxiety-Stress Disorder in Young Adults With and Without Covid-19

SUMMARY:
The purpose of this study; to examine the effects of aerobic and strength training on physical activity level, quality of life and anxiety-stress disorder in young adults with and without COVID-19. In this context, the study was planned by including 15 participants between the ages of 18-25 who had COVID-19 and 15 who did not have COVID-19. Data were collected by applying the Personal Data Form, IPAQ (International Physical Activity Form), SF-36 Quality of Life Scale, Coronavirus Anxiety Scale (CCS), Respiratory Function Tests (PFT), Six Minute Walk Test (6MWT). Aerobic training and strengthening training were applied to people with and without COVID-19 for 12 weeks. Aerobic exercise (walking) was given for 40 minutes 5 days a week, with the target heart rate being 70% of the age-corrected maximum heart rate. Strengthening exercises were applied to the upper (triceps, biceps, deltoid, pectorals) and lower (quadriceps, hamstring, gastrocnemius, tibialis anterior, hip adductors, hip flexors, hip extensors) extremities and back muscles (trapezius, latissimus dorsi) with theraband (resistance band). Significance test of the difference between two means in comparing independent group differences when parametric test assumptions are met for statistical analysis in line with the data collected from the participants; When parametric test assumptions are not met, Mann Whitney U test is used to compare independent group differences, while when parametric test assumptions are met to examine dependent group differences, the significance test of the difference between the two spouses is used; When parametric test assumptions were not met, the Wilcoxon paired two sample test was used. In all analyses, p < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Able to communicate, without hearing and/or visual impairment,
* Being between the ages of 18-25
* Not having a systemic disease
* Having had COVID-19 in the last 6 months to be included in the study group

Exclusion Criteria:

* Unable to communicate, hearing and/or visually impaired,
* Not being between the ages of 18-25
* Having a systemic disease other than COVID-19 infection,
* Having had COVID-19 more than 6 months ago.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 5 minute
  Used to define participants physical activity level
SF-36 | 10 minute
  Used to indicate the health status of participants
Coronavirus Anxiety Scale | 1 minute
  Used to evaluate experience some psychological problems such as anxiety and depression depends on COVID-19
Respiratory Function Tests | 5 minute
  Used to evaluation of the respiratory system
The 6 Minute Walk Test | 6 minute
  Used to assess aerobic capacity and endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Kücükcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If there is a reasonable request.